CLINICAL TRIAL: NCT04689451
Title: A Trial to Compare the Feasibility and Safety of Total Percutaneous Closure of Femoral Arterial Access Sites in the Veno-arterial ECMO Patients With Surgical Arterial Repair
Brief Title: Feasibility and Safety of Total Percutaneous Closure of Femoral Arterial Access Sites in the Veno-arterial ECMO Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: xuxin@GICU
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation; Myocarditis; Hypertension, Pulmonary; Pulmonary Embolism; Heart Arrest; Medication Overdoses
Keywords: decannulation; veno-arterial extracorporeal membrane oxygenation; ProGlide; vascular complications
MeSH Terms: conditions — Shock, Cardiogenic; Myocarditis; Hypertension, Pulmonary; Pulmonary Embolism; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perclose ProGlide: Perclose ProGlide group: use Perclose ProGlide to suture the artery
- Surgical Arterial Repair: Surgical Arterial Repair group : suture the artery by surgery

SUMMARY:
The most frequent access site for veno-arterial extracorporeal membrane oxygenation (VA-ECMO) is the common femoral artery (CFA), using either an open or percutaneous technique. Currently, percutaneous closure devices for femoral arterial access sites are approved for use only when a 10-F or smaller sheath has been used. However, the availability of the Perclose ProGlide (Abbott Laboratories, Chicago, IL) device has now made it possible to perform percutaneous vessel closure after using larger sheaths.The preclose technique using Perclose ProGlide, has been widely used in endovascular procedures. In a prospective randomized study, complication rates at the access site were similar in patients who underwent total percutaneous access (including percutaneous arteriotomy closure) than in those who underwent surgical cutdown and subsequent surgical closure. Total percutaneous closure of femoral arterial access sites increases patient comfort and decreases the rate of wound infections and lymphatic fistulas.[6,7] Furthermore, patients are mobilized and discharged earlier following the use of closure devices than with compression alone. Despite the above observations, no data have been published regarding percutaneous closure of femoral artery access sites in patients who have undergone VA-ECMO. In this study, we evaluated the safety and feasibility of a percutaneous closure technique using Perclose ProGlide to close the CFA access site after VA-ECMO.

ELIGIBILITY:
Inclusion Criteria:

- The study included all patients who underwent VA-ECMO and in whom Perclose ProGlide was deployed to achieve hemostasis during closure of the CFA site.

Exclusion Criteria:

* Patients were excluded if 24 hour and 30-day follow-up data regarding the access sites and other clinical outcomes were not available.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who underwent VA-ECMO
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Perclose technical success | 1day
  successful arterial closure of the CFA access site without the need for adjunctive successful arterial closure of the CFA access site without the need for adjunctive surgical or endovascular procedures.
Primary device failure | 1day
  obvious closure site bleeding after 2 Perclose ProGlides deployed, and complete device failure was defined as closure site bleeding which need surgical intervention

SECONDARY OUTCOMES:
Access-related complications | up to 24 hours after closure and during 30 days of follow-up.
  events that occurred at the arterial access site, including periprocedural bleeding equiring transfusion, acute lower limb ischemia, groin infection, device failure, arterial thrombosis, arterial dissection, pseudoaneurysm, femoral arterial stenosis, arteriovenous fistula, hematoma, and lymphocele in the periprocedural period

IPD SHARING:
Plan to Share IPD: No